CLINICAL TRIAL: NCT04485559
Title: PNOC021: A Phase I Trial Evaluating the Combination of Trametinib and Everolimus in Pediatric and Young Adult Patients With Recurrent Low-Grade Gliomas and High Grade Gliomas
Brief Title: Trametinib and Everolimus for Treatment of Pediatric and Young Adult Patients With Recurrent Gliomas (PNOC021)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Novartis Pharmaceuticals (Industry); Pediatric Brain Tumor Foundation (Unknown); The Lilabean Foundation for Pediatric Brain Cancer Research (Unknown)
Responsible Party: Principal Investigator, Sabine Mueller, MD, PhD, Principal Investigator, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 190819; NCI-2020-04097 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-07-13; First posted 2020-07-24 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Recurrent World Health Organization (WHO) Grade II Glioma; Low-grade Glioma; High Grade Glioma
Keywords: Mitogen-activated protein kinase (MAPK); phosphatidylinositol 3-kinase (PI3K); MAPK; PI3K
MeSH Terms: conditions — Glioma | interventions — Everolimus; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (trametinib, everolimus) (Experimental): Patients receive dosing per their assigned dose level. Treatment repeats every 28 days for up to 26 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Everolimus; Drug: Trametinib

INTERVENTIONS:
Drug: Everolimus — Given PO
  Other Names: 42-O-(2-Hydroxy)ethyl Rapamycin; Afinitor; Certican; RAD 001; RAD001; Votubia; Zortress
Drug: Trametinib — Given PO
  Other Names: GSK1120212; JTP-74057; MEK Inhibitor GSK1120212; Mekinist

SUMMARY:
This phase I trial studies the side effects and best dose of trametinib and everolimus in treating pediatric and young adult patients with gliomas that have come back (recurrent). Trametinib acts by targeting a protein in cells called MEK and disrupting tumor growth. Everolimus is a drug that may block another pathway in tumor cells that can help tumors grow. Giving trametinib and everolimus may work better to treat low and high grade gliomas compared to trametinib or everolimus alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the recommended phase 2 dose (RP2D) of trametinib given orally in combination with everolimus in pediatric and young adult patients with gliomas.

II. To describe the toxicity profile and define the dose limiting toxicities (DLTs) of the combination of trametinib and everolimus in pediatric and young adult patients with recurrent low-grade gliomas (LGG) or high grade glioma (HGG).

III. To characterize the pharmacokinetic profile of trametinib and everolimus when given in combination.

EXPLORATORY OBJECTIVES:

I. To describe the objective response rate and the 2-year progression-free survival (PFS) of LGGs to this therapy in the context of a phase I study.

II. To assess quality of life (QOL) and cognitive measures in pediatric and young adult patients with LGG or HGG.

III. To identify potential predictive biomarkers to targeted therapy in pediatric and young adult patients with LGGs.

IV. To assess endocrine outcomes in pediatric and young adult patients with LGGs.

V. To explore magnetic resonance (MR) quantitative measures of relative cerebral blood volume, permeability and apparent diffusion coefficient within the region of hyperintensity on T2-weighted images as markers of disease response and/or progression in comparison to institutional evaluation of disease response and/or progression and quantitative measures of tumor response as determined by central review (based upon both area and volumetric measures).

OUTLINE: This is a dose-escalation study.

Patients receive a combination of trametinib orally (PO) and everolimus in either of two dosing scheduled (continuous and intermittent). Treatment repeats every 28 days for up to 26 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, every 3 months for 1 year, then every 6 months for 5 years from the start of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed diagnosis of an LGG (WHO grade I-II) that is recurrent or progressive after prior treatment (biologic, chemotherapy or radiation therapy) or must have a histologically confirmed diagnosis of a high grade glioma (HGG) (WHO grade III-VI)

  * Participants with LGG who have had surgery alone are not eligible.
  * Participants with neurofibromatosis type 1 (NF-1) are eligible but must have available tissue per study requirements neurofibromatosis (NF) status will be collected
  * Participants with spinal cord primaries or disseminated disease are eligible
* For enrollment, snap frozen tissue (150 mg) or 10 unstained 10 um formalin-fixed, paraffin-embedded (FFPE) slides for comprehensive genomic testing or results of prior testing is required

  * If clinical comprehensive testing has already been performed, the requirement for submission of tissue may be waived after discussion and review of results with study chairs
* Participants must have evaluable disease
* Prior therapy: Participants must have received prior therapy other than surgery and must have fully recovered from the acute toxic effects of all prior chemotherapy, biologics, immunotherapy, or radiotherapy prior to entering this study

  * Myelosuppressive chemotherapy: Participants must have received their last dose of known myelosuppressive anticancer chemotherapy at least three weeks prior to study registration or at least six weeks if they had received nitrosourea. Biologic agents: Participant must have recovered from any acute toxicity potentially related to the agent and received their last dose of the biologic agent >= 7 days prior to study registration. For biologic agents that have a prolonged half-life, at least three half-lives must have elapsed prior to registration

    * Participants may have received prior treatment with a mitogen-activated extracellular signal-regulated kinase (MEK) or Mechanistic target of rapamycin (mTOR) inhibitor but must not have developed severe (grade III or IV) clinically significant toxicity. (Participants who developed grade III or IV toxicity which was not presumed by the treating physician to be medically significant should be discussed with the study chair or co-chair)
  * Monoclonal antibody treatment: Participants must have received their last dose at least four weeks prior to study registration
  * Radiation: Participants must have: had their last fraction of local irradiation to the primary tumor, craniospinal irradiation (> 24 Gy) or total body irradiation > 12 weeks prior to registration; investigators are reminded to review potentially eligible cases to confirm disease progression and avoid confusion with pseudo-progression
  * Bone marrow transplant: Participants must be: >= 6 months since allogeneic bone marrow transplant prior to registration; >= 3 months since autologous bone marrow/stem cell prior to registration
  * Corticosteroids: Participants who are receiving steroids must be on a stable or decreasing dose for at least 1 week prior to registration
* Karnofsky >= 50 for participants > 16 years of age and Lansky >= 50 for participants =< 16 years of age. Participants who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Peripheral absolute neutrophil count (ANC) >= 1000/mm^3 (unsupported)
* Platelet count >= 100,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
* Hemoglobin >= 8 m/dL (may be supported)
* International normalized ratio (INR) =< 1.5
* Creatinine clearance or radioisotope growth factor receptor (rGFR) >= 70 mL/min/1.73 m^2 or a serum creatinine based on age/gender as follows:

  * 1 to < 2 years: 0.6 (male), 0.6 (female)
  * 2 to < 6 years: 0.8 (male), 0.8 (female)
  * 6 to < 10 years: 1 (male), 1 (female)
  * 10 to < 13 years: 1.2 (male), 1.2 (female)
  * 13 to < 16 years: 1.5 (male), 1.4 (female)
  * >= 16 years: 1.7 (male), 1.4 (female)
* Bilirubin (sum of conjugated + unconjugated) =< 1.5 x upper limit of normal (ULN) for age
* Serum glutamate pyruvate transaminase (SGPT) alanine aminotransferase (ALT) =< 3 x ULN
* Serum albumin >= 2 g/dL
* Sodium, potassium, calcium and magnesium within 1.5 x institutional lower limit of normal (LLN) or ULN
* Participants must have cholesterol level < 350 mg/dL and triglycerides < 400 mg/dL before starting therapy. In case one or both of these are exceeded, the participant can only be included after initiation of appropriate lipid lowering medication and documentation of cholesterol < 350 mg/dL and triglycerides < 400mg/dl before start of therapy
* Participants with seizure disorder may be enrolled if well controlled. Participants must be on non-enzyme inducing anticonvulsants which are not excluded on study therapy
* Participants with neurological deficits should have deficits that are stable for a minimum of 1 week prior to registration
* Corrected QT (QTc) interval =< 450 msecs
* Left ventricular ejection fraction (LVEF) >= 50%
* Pulse oximeter (Ox) > 93% on room air
* Hypertension

  * Participants 3-17 years of age must have a blood pressure that is =< 95th percentile for age, height, and gender at the time of registration
  * Participants who are >= 18 years of age must have a blood pressure that is < 140/90 mm of Hg at the time of registration
* Participants must agree to use adequate contraception: The effects of trametinib and everolimus on the developing human fetus are unknown. For this reason, women of child-bearing potential and males of child fathering potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and 4 months after completion of trametinib and everolimus administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* A legal parent/guardian or participant must be able to understand, and willing to sign, a written informed consent and assent document, as appropriate per institutional guidelines

Exclusion Criteria:

* Participants who are receiving any other investigational agent for treatment of their tumor
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to everolimus or trametinib
* Participants without available tissue from prior surgery. (If clinical comprehensive testing has already been performed, the requirement for submission of tissue may be waived after discussion and review of results with study chairs)
* Participant is receiving any of the following medications within 7 days prior to enrollment (If participants require (re)initiation of these agents after enrollment and prior to start of therapy they will not be eligible to initiate study therapy):

  * Known strong inducers or inhibitors of CYP3A4/5, including enzyme inducing anti-convulsant drugs (EIACDs), grapefruit, grapefruit hybrids, pomelos, starfruit, and Seville oranges
  * Substrates of CYP3A4/5 with a narrow therapeutic index
  * Herbal preparations/medications (except for vitamins) including, but not limited to: St. John's wort, Kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, black cohosh and ginseng. Participants should stop using all herbal medications at least 7 days prior to enrollment
  * As part of the enrollment/informed consent procedures, the participant and/or legal parent or guardian will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the participant is considering a new over-the-counter medicine or herbal product
* Women of childbearing potential who are pregnant or breast-feeding

  * Female participants of childbearing potential must have a negative serum or urine pregnancy test within 72 hours of enrollment AND within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Human immunodeficiency virus (HIV) positive participants will be ineligible if HIV therapy regimen has not been stable for at least 4 weeks or there is intent to change the regimen within 8 weeks following enrollment, or if they are severely immunocompromised
* Participants with known hepatitis B or C are not eligible
* Participants with any clinically significant unrelated systemic illness (serious infectious or significant cardiac, pulmonary, hepatic or other organ dysfunction), which in the opinion of the investigator would interfere with the study procedures or results
* Participants with other factors that increase the risk of QT prolongation or arrhythmic events (e.g., heart failure, hypokalemia, family history of long QT interval syndrome) including heart failure that meets New York Heart Association (NYHA) class II or above are excluded

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-12-09 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of trametinib in combination with everolimus for both continuous and intermittent dosing schedules | Up to 28 days
  We will employ the Bayesian optimal interval (BOIN) design to find the MTD for both continuous and intermittent dosing schedules. The BOIN design is implemented in a simple way similar to the traditional 3+3 design, but is more flexible and possesses superior operating characteristics that are comparable to those of the more complex model-based designs, such as the continual reassessment method (CRM).
Incidence of adverse events for both continuous and intermittent dosing schedules | Up to 30 days after the last day of treatment
  Toxicities will be graded based on Common Terminology Criteria for Adverse Events (CTCAE) V5 .0 and followed for 30 days after last treatment or until resolution or returned to baseline values.
Dose limiting toxicities (DLTs) of the combination for both continuous and intermittent dosing schedules | Up to 28 days
  Any treatment related adverse event during the first cycle of therapy that leads to a dose reduction or results in delay of treatment > 7 days or which results in the permanent cessation of therapy will be considered dose limiting.
Recommended phase 2 dose (RP2D) | Up to 28 days
  The RP2D rate is selected based on isotonic regression as specified in Liu and Yuan (2015). This computation is implemented by the shiny app "BOIN" available at http://www.trialdesign.org. Specifically, select as the RP2D the dose for which the isotonic estimate of the toxicity rate is closest to the target toxicity rate.
Maximum Concentration (Cmax) of trametinib and everolimus | Up to 5 years
  Plasma trametinib and everolimus concentration-time data will be analyzed using a classic non-compartmental approach and/or population-based compartmental methods using non-linear mixed effects modeling. Individual pharmacokinetic parameters of interest after single and repeated doses (i.e., maximum plasma concentration Cmax from 0 to 24h will be calculated from the pharmacokinetic model. Trametinib and everolimus pharmacokinetics after single dose will be compared to trametinib and everolimus pharmacokinetics after repeated doses.
Area Under the Curve (AUC) of trametinib and everolimus | Up to 5 years
  Plasma trametinib and everolimus concentration-time data will be analyzed using a classic non-compartmental approach and/or population-based compartmental methods using non-linear mixed effects modeling. Individual pharmacokinetic parameters of interest after single and repeated doses (i.e., area under the curve from 0 to 24h will be calculated from the pharmacokinetic model. Trametinib and everolimus pharmacokinetics after single dose will be compared to trametinib and everolimus pharmacokinetics after repeated doses.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Mueller, Principal Investigator — University of California, San Francisco
Locations (18):
- United States (18):
  - University of Alabama at Birmingham, Children's of Alabama, Birmingham, Alabama
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California, San Diego Rady Children's Hospital, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - John Hopkins University, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Children's Minnesota, Minneapolis, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - Joseph M. Sanzari Children's Hospital at Hackensack University Medical Center, Hackensack, New Jersey
  - New York University, New York, New York
  - Doernbecher Children's Hospital Oregon Health & Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University Of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No